CLINICAL TRIAL: NCT01622153
Title: A Prospective Study and Clinical Evaluation of Pre & Post Operative Treatment Comparison of Electrical and Formocresol Pulpotomy Procedures in Primary Molars of Children Undergoing General Anesthesia
Brief Title: Electrical and Formocresol Pulpotomy in Primary Molars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Use of Formocresol for pulpotomies ws discontinued.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Gerald Feretti, DDS, MS, MPH, Chair of Pediatric Dentistry, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021117
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Reversible Pulpitis; Caries
MeSH Terms: interventions — Electrosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formocresol (control) (Placebo Comparator): This will consist of patients who are ASA I or II status, 3-8 years old, males and females, and present with restorable primary molars with reversible pulpitis and free of clinical radiographic signs of pulp pathology. From these study participants, they will be randomly assigned to this or other group. Patients in this group will receive a pulpotomy. Cotton pellets are saturated with conventional 1:5 dilution of Buckley's formocresol into the canal orifice for 5 minutes for complete hemostasis. IRM (Zinc Oxide Eugenol) cement will then be placed to seal the pulp chamber. A stainless steel crown will be cemented with Ketac Cement that was triturated for 10 seconds to complete the pulpotomy procedure and final restoration.
  Interventions: Procedure: Formocresol application after pulpotomy preparation
- Laser (Active Comparator): This will consist of patients who are ASA I or II status, 3-8 years old, males and females, and present with restorable primary molars with reversible pulpitis and free of clinical radiographic signs of pulp pathology. From these study participants, they will be randomly assigned to this or other group. Patients in this group will receive a pulpotomy. Then a GENTLEray 980 Soft Tissue diode laser (Power: 3.0W, Mode: PW, Fiber: 300µm, Ton: 100ms, Toff: 100ms, Timer: cont) will be used to vaporize the residual pulp tissue and complete hemostasis. IRM (Zinc Oxide Eugenol) cement is then placed to seal the pulp chamber. A stainless steel crown cemented with Ketac Cement for the full coverage final restoration completes the pulpotomy procedure.
  Interventions: Procedure: GENTLEray 980 Soft Tissue diode laser

INTERVENTIONS:
Procedure: Formocresol application after pulpotomy preparation — 1:5 Buckley's Formocresol dilution applied for 5 minutes or until hemostasis achieved
  Other Names: Buckley's solution, baby root canal, primary root canal
  Arms: Formocresol (control)
Procedure: GENTLEray 980 Soft Tissue diode laser — Application to pulp chamber until hemostasis achieved
  Other Names: soft tissue laser, electrosurgery, baby root canal
  Arms: Laser

SUMMARY:
1. The investigator hypothesize that the Laser pulpotomy will provide adequate and comparable success clinically in primary molars.
2. The investigators hypothesize that the Laser pulpotomy will provide adequate and comparable success radiographically in primary molars.

DETAILED DESCRIPTION:
The health of teeth, their supporting tissues and maintaining their integrity is the primary goal of pulp therapy. Conservative pulp therapy for primary teeth aims to maintain pulp vitality, reduce the need for a pulpectomy, and promote the integrity and retention of such teeth until appropriate exfoliation.(51) A pulpotomy is usually performed for carious exposures of primary teeth with normal pulp or reversible coronal pulpitis, or primary teeth pulpally exposed by trauma (AAPD 2009). A pulpotomy requires healthy radicular pulp capable of healing after amputation of inflamed or infected coronal pulp [Fuks and Eidelman, 1991]. After the coronal pulp is amputated, the remaining vital radicular pulp tissue surface is treated with a long-term clinically successful medicament such as Buckley's Solution of formocresol. (46-52) Electrosurgery has also demonstrated success. (53) The coronal pulp chamber is filled with zinc/oxide, eugenol, or other suitable base, and the tooth is restored with a restoration that seals the tooth from microleakage. The most effective long-term restoration has been shown to be a stainless steel crown.

When the coronal tissue is amputated, the remaining radicular tissue is judged to be vital without suppuration, purulence, necrosis, or excessive hemorrhage that cannot be controlled with a damp cotton pellet after several minutes. In addition to this, if there are no radiographic signs of infection or pathologic resorption then a pulpotomy procedure is indicated. (Camp JH, Fuks AB) Despite concerns of toxicity, mutagenicity and carcinogenicity [Swenberg et al., 1980; Goldmacher and Thilly, 1983; Ranly and Horn, 1987], formocresol (FC) remains a commonly used primary tooth pulpotomy medicament [Hingston et al., 2007]. Various clinical and radiographic success rates (59-100%) have been reported [Mejare, 1979; Naik and Hegde, 2005], attributed to intra-patient variations, clinician and assessor factors, FC concentrations and application times, coronal seal, and study durations.

As technology continues to improve, it allows dentists to treat patients with greater precision, meaning less pain and quicker healing. The diode laser is used in many different dental procedures. It is most commonly used to perform soft-tissue surgery in the mouth. The diode laser's high-energy beam kills bacteria, thus it is often used to sterilize areas of the mouth before or during root canal procedures. (Laser-dentistry/diode-laser) The diode laser represents a whole new way of thinking about dental care. Laser treatment is less painful, more convenient, and more effective than many traditional dental treatments. A study by Bahrololoomi Z, Moeintaghavi A, comparing FC and electrosurgery pulpotomy after nine months of follow up found that clinical and radiographical success rates were 96% and 84% respectively in the electrosurgical group and 100% and 96.8% respectively in the formocresol group. There was no statistical significance and the results showed that the failure rates for electrosurgery pulpotomy were equal to those of formocresol pulpotomy.

Purpose:

Dental care has recently been identified as the most prevalent unmet health need amongst US children (AAPD 2009). This research study investigates another treatment method to help provide dental care to these children by evaluating the success rate of a laser (electrical) pulpotomy compared to formocresol pulpotomy in primary molars with carious pulp exposure. There is a need to study and assess the laser pulpotomy method in order to help create a more efficient and painless treatment.

Study Design and Procedures:

We will perform a prospective study and clinical evaluation of patients ranging from ages 3-8 years old treated under general anesthesia from June, 2010 to June, 2014. The review and analysis will be completed over a four year time period. The patients participating in this study will include those presenting themselves as patients to the Tapper Pediatric Dentistry clinic at Rainbow Babies Children's Hospital. These patients will only be scheduled to be treated in the operating room when it is indicated as the best treatment option. Treatment under General Anesthesia is indicated when: 1. Patient is uncooperative due to a lack of psychological or emotional maturity and/or mental, physical, or medical disability. 2. Patients for whom local anesthesia is ineffective because of acute infection, anatomic variations, or allergy. 3. Extremely uncooperative, fearful, anxious, or uncommunicative child or adolescent. 4. Patients requiring significant surgical procedures. 5. Patients for whom the use of GA may protect the developing psyche and/or reduce medical risk. 6. Patients requiring immediate, comprehensive oral/dental care (AAPD 2009). The patients will then be consented and informed on the same day of the OR appointment. They will be given specific post-op instructions both verbally and in written form. They will be scheduled for a two-week follow-up appointment in the clinic following dental treatment. Informed consent must be obtained by the parent/guardian of the patients that will participate in the study and receive pulpotomy treatment with the laser technique. Other patients, regardless of the study, will have pulpotomy treatment using the traditional formocresol technique.

All patients will receive general endotracheal anesthesia while receiving comprehensive dental treatment. General anesthesia will be provided using a combination of inhaled anesthetics and propofol intravenously. General anesthesia will be supplemented with intravenous opioid analgesics, ketorolac unless contraindicated, and anti-mimetics. The anesthetic approach will not be influenced by participation or non-participation of patients in the study.

The patient's name, date of birth, and medical history will be obtained from each patient chart. This PHI will be utilized to keep track of patient demographics for the study. Patients scheduled for the operating room will be seen for a post-op two week follow up appointment and regular dental visits regardless of whether or not they are participating in the study.

Of the eligible subjects a randomized clinical trial will be performed on 90 primary molars in children aged 3-8 years. Two preoperative bite wing radiographs will be taken. The teeth will be treated for pulp therapy using either a conventional formocresol (30 controls and 30 study teeth) or GENTLEray 980 Soft Tissue diode laser (30 study teeth) technique. 30 Controls: The procedure for these 30 subjects is conducted using a #8 round diamond bur to remove occlusal tooth structure for pulp chamber access and removal of coronal pulp. Cotton pellets are saturated with conventional 1:5 dilution of Buckley's formocresol into the canal orifice for 5 minutes for complete hemostasis. After this, a Chlorhexidine Gluconate 0.12% rinse will be applied to decrease the bacterial level. Then, placement of 35% Phosphoric Acid Etch for 15-30 seconds is rinsed off and dried until the tooth has a white, chalky appearance. One layer of Optibond Solo is placed into the pulp chamber and light cured for 10 seconds with a 3M ESPE Elipar S10 light curing device. IRM (Zinc Oxide Eugenol) cement will then be placed to seal the pulp chamber. A stainless steel crown will be cemented with Ketac Cement that was triturated for 10 seconds to complete the pulpotomy procedure and final restoration. 30 Conventional Formocresol: The procedure for these 30 subjects is conducted using a #8 round diamond bur to remove occlusal tooth structure for pulp chamber access and removal of coronal pulp. Cotton pellets are saturated with conventional 1:5 dilution of Buckley's formocresol into the canal orifice for 5 minutes for complete hemostasis. After this, a Chlorhexidine Gluconate 0.12% rinse will be applied to decrease the bacterial level. Then, placement of 35% Phosphoric Acid Etch for 15-30 seconds is rinsed off and dried until the tooth has a white, chalky appearance. One layer of Optibond Solo is placed into the pulp chamber and light cured for 10 seconds with a 3M ESPE Elipar S10 light curing device. Dyract compomer will then be placed to seal the pulp chamber. A stainless steel crown is cemented with Ketac Cement that was triturated for 10 seconds to complete the pulpotomy procedure and final restoration. 30 Laser Diode: The procedure for these 30 subjects is conducted using a #8 round diamond bur to remove occlusal tooth structure for pulp chamber access and removal of coronal pulp. Then a GENTLEray 980 Soft Tissue diode laser (Power: 3.0W, Mode: PW, Fiber: 300µm, Ton: 100ms, Toff: 100ms, Timer: cont) will be used to vaporize the residual pulp tissue and complete hemostasis. After completion of hemostasis, a Chlorhexidine Gluconate 0.12% rinse will be applied to decrease the bacterial presence. Subjects will then receive placement of 35% Phosphoric Acid Etch for 15-30 seconds followed by 10 second light cured optibond solo. IRM (Zinc Oxide Eugenol) cement is then placed to seal the pulp chamber. A stainless steel crown cemented with Ketac Cement for the full coverage final restoration completes the pulpotomy procedure.

Following the pulpotomy procedures, the teeth will be evaluated for clinical and radiographic success at 6 months post-op and 12 months post-op appointments at the Tapper Pediatric Dental Clinic at Rainbow Babies Children's Hospital. The study teeth treated will be evaluated clinically based on the presence of the following: (1) pain (2) abscess (3) mobility. Radiographic success will be determined by evaluating a bite wing x-ray taken at the two post-op appointments for the presence of the following: (1) internal resorption (2) external resorption and (3) furcation radiolucency.

Risks:

The only physical risk in laser therapy is the risk of eye damage. While eye damage has not been reported to date, we must still consider it as a possible risk. Because these study subjects will be under General Anesthesia their eyes will already be closed and covered. Suitable protective goggles should be worn by the investigator and assistants. Other possible risks associated with this study include risks from anesthesia- (Nausea, vomiting, epistaxis, fever, discomfort/pain). There are minimal to no risks involved in this research study.

Benefits:

Pulpotomy treatment maintains the vitality of the tooth as well as the supporting tissues. The longevity and prognosis of having a laser pulpotomy versus a formocresol pulpotomy treatment has been considered to be just as beneficial. Through this research study, we can further prove this new finding. Maintaining your primary dentition is extremely important and this study will provide insight on how advances in dental technology can help better treat carious teeth in more efficient and painless ways.

Alternatives:

Due to the nature of this research the only alternative is to not participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Restorable carious primary molars with reversible pulpitis and free of clinical or radiographic signs of pulp pathology
2. Males and females
3. Children ages 3-8 years old
4. Children classified under ASA I or II status

Exclusion Criteria:

1. Excluded will be primary molars with clinical or radiographic signs of pathology
2. Children not within age range
3. Absence of parent/caregiver
4. Mentally disabled parent/caregiver
5. Patients not returning for 6 month and 12 month follow up examination appointment

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Radiographic | 6, 12, and 18 months
  Failure is identified as radiographic: furcation radiolucency, external root resorption

SECONDARY OUTCOMES:
Clinical | 6, 12, 18 months
  Failure determined by clinical presence of: mobility, abscess, spontaneous pain, suppuration

CONTACTS AND LOCATIONS:
Overall Officials: Gerald A Ferretti, DDS, MS, MPH, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospital-Rainbow Babies & Children's Hospital, Cleveland, Ohio, United States